CLINICAL TRIAL: NCT06303674
Title: Effects of Brain Breaks on Educational Achievement in Children With and Without ADHD: The Break4Brain Project
Brief Title: Effects of Brain Breaks on Educational Achievement in Laboratory Settings: The Break4Brain Project
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government); European Regional Development Fund (Other); State Research Agency, Spain (Other Government)
Responsible Party: Principal Investigator, Josep1, Senior Lecturer, University of the Balearic Islands
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 301CER22; PID2021-123357OA-I00 (Other Grant/Funding Number: Ministry of Science and Innovation - Spanish State Research Agency - European Regional Development Fund)
Record Dates: First submitted 2024-02-01; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: ADHD
Keywords: brain breaks; exercise; brain function; executive function; academic performance
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The design of the study is a within-participants crossover pretest-posttest comparison design under laboratory settings will be used. In this design, all participants will engage in all experimental conditions (on separate days), with the order of the experimental conditions being counterbalanced across participants and outcomes assessed following each experimental condition.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical activity with engaging cognitively (Experimental): This experimental condition involves engaging in physical activity interspersed with rest periods based on cognitive tasks.
  Interventions: Behavioral: Physical activity with engaging cognitively
- Physical activity without engaging cognitively (Experimental): This experimental condition involves engaging in physical activity interspersed with rest periods (without cognitive tasks).
  Interventions: Behavioral: Physical activity without engaging cognitively
- Cognitively engaging control conditions (No Intervention): In this condition, participants will be suggested to watch a video while seating/resting for 10 minutes.

INTERVENTIONS:
Behavioral: Physical activity with engaging cognitively — This experimental condition will follow the following structure: involving 10 consecutive, 30 second-blocks of physical activity. This experimental condition will focus on aerobic metabolism. The total exercise time commitment is 10 minutes (30 seconds of working - 30 seconds of executing an engaging cognitive task, 1:1 work-to-rest ratio), plus 5 minutes of warm-ups and 5 minutes of cool-down activities. The cognitive task consists of solving various "tangrams".
  Arms: Physical activity with engaging cognitively
Behavioral: Physical activity without engaging cognitively — This experimental condition will replicate the structure of the preceding one. Participants will engage in physical activity, guided by video observation and imitation. However, during the rest periods, they will refrain from engaging in cognitive tasks
  Arms: Physical activity without engaging cognitively

SUMMARY:
Advancement in teaching methods, together with the frenetic change in the lifestyles of the school population, provides a unique opportunity to advance scientific knowledge. The current project, called "The Break4Brain Project", aims to examine the acute (transient) effects of physical activity on brain function, cognition, and academic performance in children with and without Attention Deficit Hyperactivity Disorder (ADHD). Specifically, a total of 60 children between 10 and 12 years old will be included with (n=30) and without (n=30) ADHD. The study will use an intra-subject design of isolated conditions with four measurement moments where the children will perform three different experimental conditions lasting 10 minutes, which will be randomized in a counterbalanced manner. These experimental conditions will be based on physical activity engaging cognitively, physical activity without engaging cognitively, and cognitively engaging control condition. This project could have a significant impact in the educational field, since, if brain function, cognition, and academic performance prove to be favorably stimulated, acutely, by physical activity through active breaks, these could be prescribed as an effective teaching strategy for children with and without ADHD in the school setting.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 10-12 years diagnosed with ADHD by a recognized diagnostic procedure.
* Children aged 10-12 years without any neurodevelopmental impairment.

Exclusion Criteria:

* Children who have serious physical or mental disorders.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Academic achievement | 4 times (during 4 weeks)
  In this research, only the general academic fluency index was administered, consisting of the reading, mathematics, and writing fluency subtests. Reading fluency assessed the participant's capacity to read simple sentences rapidly, mathematical fluency gauged the ability to quickly solve simple addition, subtraction, and multiplication problems, and writing fluency measured the skill to formulate and write sentences promptly.
Inhibition | 4 times (during 4 weeks)
  Flanker Test: Assessed inhibitory control of irrelevant stimuli. Congruent stimuli facilitated processing, while incongruent ones hindered it.
Working memory | 4 times (during 4 weeks)
  n-back Test: Evaluated working memory's information updating. Participants matched stimuli to the one 'n' items ago, with increasing difficulty.
Sustained attention | 4 times (during 4 weeks)
  Conners CPT-3 Attention Test: Examined sustained attention with 360 trials, 18 blocks, and varying intervals. 90% featured non-X target stimuli. Assessment included scaled scores for attentional capacity (d'), error categorization, and reaction metrics.
Brain function | 4 times (during 4 weeks)
  Event-related brain potentials (ERPs), acquired from the electroencephalogram, served as a metric for brain response to discrete events. Neuroelectric activity was captured from 14 scalp electrode sites, arranged using the EMOTIV EPOC X and its corresponding software. Selected components of event-related brain potentials were assessed, with a focus on analyzing the amplitude and latency of P3 (also referred to as P300). A higher P3 amplitude was considered indicative of an enhanced ability to enlist attentional resources, while a lower P3 latency was considered indicative of heightened cognitive processing speed. In study I, ERPs were concurrently recorded during cognitive function (not CPT-3).

SECONDARY OUTCOMES:
Physical fitness and body composition | baseline
  Were measured using the ALPHA Physical Fitness Test Battery.
Physical activity levels and sleep | baseline
  Were assessed using Actigraph wGT3X-BT accelerometers, which participants carried throughout their four-week involvement in the project. Additionally, sedentary lifestyle levels were gauged using the Youth Activity Profile (YAP).
Self-reported sedentary patterns | baseline
  Sedentary lifestyle levels were also gauged using the Youth Activity Profile (YAP).
Motor proficiency | baseline
  Was assessed using the Bruininks-Oseretsky Test of Motor Proficiency.
Biological maturation | baseline
  Was measured using maximum height velocity (PHV), an indicator reflecting the peak velocity of height growth during childhood. Weight, height, and sitting height were utilized to calculate VPM based on Moore's equations.
ADHD symptoms | baseline
  Was evaluated utilizing the Conners Scales 3-Parent Version.
IQ | baseline
  Was assessed using the Kaufmann Brief Intelligence Test (K-BIT).
Socioeconomic levels | baseline
  The parents' socioeconomic status was determined using the Family Affluence Scale-II.
Educational levels | baseline
  The parents' educational level was determined using a custom questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Adrià Muntaner-Mas, PhD, Principal Investigator — University of the Balearic Islands
Locations (1):
- University of the Balearic Islands, Palma, Balearic Islands, Spain